CLINICAL TRIAL: NCT06390605
Title: a Non-invasive Ultrasonographic Method for the Measurement of Intra-abdominal Pressure in Combination With External Pressure
Brief Title: a Ultrasonographic Measurement of Intra-abdominal Pressure
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZWQ21886-2024-1
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Critical Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intra-abdominal pressure (IAP) refers to the stable pressure in a closed cavity. Its magnitude is determined by the compliance of the abdominal wall and the pressure of the abdominal cavity contents, and it increases with inhalation and decreases with exhalation. Due to fluid retention, organ failure, use of ventilators, and other reasons, critically ill patients have higher intra-abdominal pressure, ranging from 5-7mmHg. However, the expansion capacity of the peritoneal cavity is limited. As the internal pressure rises, when the intra-abdominal pressure rises above 12 mmHg, intra-abdominal hypertension (IAH) occurs. Elevated IAP has harmful physiological effects on almost all organ systems, including the central nervous system, cardiovascular, respiratory, kidney, gastrointestinal, and liver systems. When IAP continues to rise and is accompanied by new or progressive organ failure, it develops into abdominal compartment syndrome (ACS), which is the end-stage manifestation of severe IAH.

Currently, there are various methods for measuring intra-abdominal pressure, including direct intraperitoneal measurement, transbladder measurement, gastric measurement, superior and inferior vena cava measurement, rectal measurement, and noninvasive measurement. However, the most commonly used clinical method is indirect transbladder measurement. This technique is clinically feasible and accurate, making it the internationally recognized "gold standard" for intra-abdominal pressure monitoring. Nevertheless, it has been reported that the accuracy and reproducibility of intra-bladder pressure measurements can be influenced by many factors, resulting in a large coefficient of variation in intra-abdominal pressure measurements obtained by this method. Additionally, the indirect transbladder measurement technique is cumbersome, discontinuous, and carries a potential risk of infection. Therefore, the development of noninvasive, safe, and reliable IAP monitoring techniques or methods has garnered widespread attention from scholars both domestically and internationally.

This study measures IAP using a combination of ultrasound and external pressure application. By comparing it with the gold standard, intra-bladder pressure measurement, we observe the accuracy and reliability of this measurement method. The aim is to provide a noninvasive, fast, accurate, and reliable method for measuring intra-abdominal pressure in critically ill patients.

DETAILED DESCRIPTION:
1. Design and Manufacture of a Device for Measuring Pressure Applied by Ultrasonic Probe

   Four pressure-sensing patches, each with a diameter of 0.5mm, are placed at the four corners of the linear array probe. The placement positions are based on not affecting ultrasonic imaging, and they are fixed around the probe through a bracket. The wires of the four pressure-sensing patches are connected to a pressure measurement module, which can process the pressure exerted on the four patches and calculate the average pressure. Finally, the pressure exerted on the four patches and the average pressure value are displayed on the monitor.
2. Measurement of IAP Using Ultrasound Combined with External Pressure Application

   The operation was performed by two researchers who were unaware of each other's measurement results. The first researcher had more than 3 years of experience in critical ultrasound operation and was familiar with the ultrasound combined with external pressure application method and operation procedure before the study began, so no additional training was required. The second researcher also had more than 3 years of experience in critical ultrasound operation but was not aware of the ultrasound combined with external pressure application method. The first researcher trained the second researcher, only informing the latter of how to use ultrasound combined with external pressure to measure intra-abdominal pressure. Using a Philips ultrasound system (model: IU22) and a linear array probe (frequency: 5-12 mHz), preset superficial parameters and two-dimensional mode were selected. The researchers adjusted the depth and gain to clearly display the peritoneal line, with the focus centered on the peritoneal line and the grayscale compression set to automatic adjustment mode, generally between 60% and 70%.

   During measurement, the patient lies on their back with the abdominal wall relaxed. The bladder is emptied through a urinary catheter. The measurement device for pressure applied by the ultrasonic probe is fixed to the probe and gently placed 2cm above the navel, perpendicular to the abdominal wall. Observe and record the original shape of the peritoneal line, then gradually apply pressure until the peritoneal line changes shape towards the peritoneal cavity and record the pressure value. Finally, quickly remove the pressure on the probe and observe whether the peritoneal line returns to its original shape. If the peritoneal line returns to its original shape, the recorded pressure value is the intra-abdominal pressure. Each researcher measures twice consecutively, and the average value is taken as the final value. Each patient is measured once within 24 hours of ICU admission and again after 72 hours.
3. Measurement of IAP by Intra-bladder Pressure Method

After the measurement using ultrasound combined with external pressure, a third researcher who is unaware of the ultrasound measurement results performs the intravesical pressure method. This is done according to the standards recommended by the World Abdominal Compartment Syndrome Federation. The specific method is as follows: insert a urinary catheter into the bladder, empty the urine from the bladder, and then inject 25ml of normal saline into the bladder through the catheter. Connect a T-junction and a pressure measuring tube. During the measurement, the patient lies on their back with the abdominal covering removed, using the axillary midline as the "zero" point. The height of the water column represents the intra-abdominal pressure. During the measurement process, the patient should maintain calm breathing, and the reading should be taken at the end of exhalation to minimize errors. If the patient is using a ventilator with positive end-expiratory pressure, the ventilator tubing should be disconnected for measurement to reduce the influence of ventilator-assisted ventilation on intra-abdominal pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indwelling catheters who can undergo intra-bladder pressure measurement.
* Patients suspected of having elevated intra-abdominal pressure.
* Patients who have agreed to participate in this study and signed a written informed consent form, either by themselves or through their immediate family members.

Exclusion Criteria:

* Patients with wounds in the middle of the abdominal wall, making it impossible to perform abdominal wall pressure measurements.
* Patients with pathological changes in the abdominal wall, such as congenital malformations, injuries, hematomas within the rectus sheath, infections, tumors, hernias, etc.
* Patients whose water column does not show respiratory phase changes during intra-bladder pressure measurement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill patients admitted to a tertiary hospitals in Shanghai, China from May 2024 to April 2025
Sampling Method: Non-Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Pearson correlation coefficient | From May 2024 to April 2025
  Pearson correlation coefficient between golden standard and ultrasonographic method

CONTACTS AND LOCATIONS:
Overall Officials: weiqing zhang, Ph.D., Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided